CLINICAL TRIAL: NCT03836430
Title: The Impact of a Newborn Behavioral Intervention on the Mental Health of Mothers With Late Pre-Term Infants
Acronym: BabyAMOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Child Trends (Other)
Responsible Party: Principal Investigator, Lise Carolyn Johnson, Pediatrician, Department of Pediatric Newborn Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018P001771
Record Dates: First submitted 2019-02-05; First posted 2019-02-11 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Postpartum Depression; Preterm Infant; Infant Development
Keywords: newborn behavioral observation; late preterm; postpartum depression
MeSH Terms: conditions — Depression, Postpartum; Premature Birth

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment involving two groups of participants. Group A received the intervention of Newborn Behavior Observation (NBO) sessions and Group B did not.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newborn Behavioral Observation (Experimental): The Newborn Behavioral Observation-Family Wellness (NBO-FW) intervention is the experimental arm of this RCT. It consists of 3 NBOs - 2 during the birth hospitalization and the third at 6 weeks post-discharge as well as a journal with prompts for mothers to reflect on their infant's behavior and their own transition to motherhood. NBOs are clinical relationship-building tools used by trained clinicians/therapists to help parents understand their babies' unique language.
  Interventions: Behavioral: Newborn Behavioral Observation-Family Wellness (NBO-FW)
- Usual care (No Intervention): This arm is the usual care arm. Of note, both arms receive 2 parenting books, one at hospital discharge and one at 6 weeks post-discharge.

INTERVENTIONS:
Behavioral: Newborn Behavioral Observation-Family Wellness (NBO-FW) — The intervention has been described in the arm description.
  Arms: Newborn Behavioral Observation

SUMMARY:
Preterm birth is a serious public health issue, affecting 10% of all births in the US alone. Three quarters of these infants are born between 34 0/7 and 36 6⁄7 weeks' gestation or late-preterm (LP). Mothers of LP infants are at increased risk for postpartum stress, depression and mother-infant interaction problems posing significant risks for infant development. Our proposed project will advance the fields of maternal and child health by examining the impact of the Newborn Behavioral Observations Family Wellness (NBO-FW), a dyadic, two generational intervention targeting maternal wellbeing and early mother-infant relations in families of LP born infants. The NBO-FW is a 12week preventative intervention aimed at promoting maternal mental health and positive parenting. It is based on the highly successful NBO intervention developed by our team and applied across five continents, but with important new elements targeting maternal mental health and the needs of high-risk LP infants and their families. Participants will consist of 200 first-time mothers and their LP infants (100 intervention and 100 control dyads) born at Brigham and Women's Hospital (BWH), an urban teaching hospital of Harvard Medical School and the largest maternity care provider in Boston. Data will be collected at three time points: during the birth hospitalization, at a follow-up visit at 4-6 weeks corrected gestational age, and at a further visit 10-12 weeks after birth. Outcomes will include standardized measures of maternal stress, depression, parenting confidence, and observed mother-infant interaction. Information about infant health care practices and maternal/infant health will also be recorded. We hypothesize that, compared to mothers in the care as usual control group, first-time mothers of LP infants who receive the NBO-FW will demonstrate a) lower levels of stress and depression, b) greater parenting confidence, c) higher quality interactions with their infants (e.g., positive affect, sensitivity, responsiveness, emotional connection); and (d) engage in more optimal infant health care practices.

DETAILED DESCRIPTION:
Preterm birth is a serious public health issue, affecting 10% of births in the US alone. The vast majority of these infants are born between 32 and 37 weeks of gestation and are at increased risk of neurodevelopmental problems. The mothers of these infants are also at increased risk for postpartum stress, depression and mother-infant interaction problems which can further exacerbate child risks. Specific maternal and family challenges include mother-infant emotional disconnection, less sensitive maternal care behavior, and reduced engagement in healthy infant care practices such as breastfeeding.

To date, relatively little attention has been given to addressing the needs of preterm born (>32 and <37 weeks of gestation) infants and their families, with most research focusing on the very and extremely preterm born infant. As a result, there are few to no interventions that specifically: a) address the needs of the preterm infant and their caregivers; b) offer parent education; c) foster a close mother-infant relationship; and d) seek to provide support and empowerment of mothers. This stands in contrast to an extensive body of experimental and human infant research showing that early mother-infant contact is essential for both maternal wellbeing and offspring development, with disruptions to this early relationship having lifelong negative effects for the infant.

This research project meets this important gap, with the goal of advancing the fields of maternal and child health by examining the impact of a dyadic two-generation, Newborn Behavioral Observations-Family Wellness (NBO-FW) intervention on early maternal wellbeing and mother-infant relations in families of preterm born infants.

There is now good evidence to support the importance of early intervention as a preventative strategy to reduce the risks of longer term development problems in both typically developing and high-risk populations of mothers and infants. Intervening early with young children who are at risk for developmental delay has been shown to positively impact children's developmental outcomes across multiple functional domains, spanning health, language, cognitive and social-emotional development. In addition, families benefit from early intervention because it can increase their ability to understand and meet their child's needs, as well as mitigate stressors that may be adversely impacting maternal wellbeing, the mother-infant relationship and in turn, healthy child development.

Original Newborn Behavioral Observation Intervention The original NBO developed here in Boston by Kevin Nugent and colleagues is an interactive observational tool used by clinicians to strengthen the relationship between parents and infants from birth to age 3 months, or even longer in the case of the at-risk infant. As such, it is a flexible, short-term, family-centered early intervention strategy that is suitable for use and widely used in newborn units, the Neonatal Intensive Care Unit (NICU), obstetric, pediatric, and other primary care settings.

During an NBO session, a certified clinician and parent observe the newborn together for about 15-20 minutes. The focus is on 18 neurobehavioral items designed to capture the infant's visual, auditory, and perceptual abilities used by the infant to explore their world and engage in mutually responsive face-to-face interaction. These items include observations of the infant's capacity to habituate to external light and sound stimuli (sleep protection); the quality of motor tone and activity level; the capacity for self-regulation (including crying and consolability); response to stress (indices of the infant's threshold for stimulation such as color change, startles and tremors); and the infant's visual, auditory, and social-interactive capacities (degree of alertness and response to both human and non-human stimuli). The original NBO is now used widely as a clinical tool throughout Europe, Australasia, Asia, Africa, and North America.

Existing data from evaluations of the NBO dyadic intervention demonstrate positive impacts on both maternal postpartum depression risk and the quality of mother-child interactions in depressed mothers and preterm infants hospitalized in the NICU. Although it's effectiveness with first-time mothers and their late preterm infants has not been evaluated, there is some support for its utility. Specifically, Nugent and Bartlett have conducted a randomized controlled trial (RCT) with first-time mothers and their full-term born infants (n = 106) in hospital and home settings. They found that the NBO was associated with a 75% reduction in maternal symptoms of depression one month after birth. A second smaller RCT study by the same authors (n = 35) with mothers and their full-term infants, also showed that mothers who received an NBO intervention were 2.5 times more likely to be rated as sensitive caregivers than non-intervention control mothers. Their infants were also observed, in turn, to be 2.8 times more responsive to their mothers, suggesting a stronger mother-infant connection. Finally, the NBO has been linked with increased maternal parenting confidence, enhanced interactions between mothers and their high-risk newborns, and increased parental knowledge of infant behaviors and competencies across a range of high risk populations.

Our Enhanced Newborn Behavioral Observation - Family Wellness (NBO-FW) Intervention:

In collaboration with Nugent and Bartlett, we have developed an extended NBO intervention. This new intervention termed the Newborn Behavioral Observation - Family Wellness (NBO-FW) approach builds on the strengths of the NBO but includes additional resources and strategies to promote parental wellbeing and mental health, as well as greater parental self-reflection on their infant and themselves as parents aimed at helping new mothers of a preterm born infant bond with their baby, feel better about themselves, and to be a more confident and competent parent.

This new NBO-FW approach is a 12-week preventative intervention that will consist of 1-2 in-person NBO-FW session in the hospital followed by a tele-health follow-up visit and a third outpatient in-person NBO-FW session with a trained and NBO certified therapist. These visits will be supplemented by the use of a parental self-reflection guide between sessions to maintain maternal engagement in the intervention and to further foster the dyads progress in understanding each other. All therapy sessions will be completed by an appropriately qualified mental health/early intervention professional trained and supervised by Kevin Nugent and Lise Johnson.

Against this background, the overall objective of this research project is to examine whether the Newborn Behavioral Observations-Family Wellness (NBO-FW) intervention leads to better maternal mental health, healthier mother-infant interactions, parenting confidence, and better infant health care practices in new mothers giving birth to a preterm born infant.

The proposed project aims to advance understanding of how to intervene successfully to improve postpartum maternal mental health, parent-child relations, and mothers' infant health care practices in high risk families. The strategy, methodology, and data analyses used to accomplish these aims are based on evidence generated from the first RCT studies conducted by Drs. Nugent, Bartlett, and colleagues. As such, the NBO-FW intervention has the potential to fulfill an important unmet need in supporting parents and their high-risk newborns in the early days and weeks of life. Potential benefits to patients will include additional assessments of their infant's health and wellbeing, as well as additional individualized support in hospital and during their transition to home. More broadly, study findings will advance knowledge about how best to improve outcomes for future preterm infants and families.

There are multiple strengths and unique qualities of the NBO-FW intervention that support its chances of research and clinical success. These include:

* Positive adaptive model. Rather than being based on a deficit model of illness, the NBO-FW is based on a positive adaptive developmental model that has been shown across a number of studies to help mothers learn to understand and care for their newborns.
* Critical time of opportunity. The birth of a child is one of the most important normative crises of life. New mothers may be uniquely open to change and support in the first days and weeks in ways that do not necessarily persist once the adjustments - positive or negative - to life with their new baby have been made and caregiving patterns are established. Appropriate for use within the first days following birth, the NBO-FW leverages this opportunity to its greatest potential.
* Efficient, short term intervention timed to coincide with routine medical care. The NBO-FW intervention is an efficient, cost-effective tool for addressing the common condition of postpartum stress and depression, as well as fostering positive parenting and infant health care practices. The NBO-FW intervention can be completed with a limited number of encounters over the first 4-6 weeks of life and is designed so that it can be implemented in tandem alongside routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* First time mothers of singleton newborns born between 32 and 37 weeks of gestation
* Mother fluent in either English or Spanish

Exclusion Criteria:

* Maternal history of major psychosis or suicidality
* Mother currently addicted to drugs or alcohol or being treated for drug addiction
* Health condition limiting mother's ability to care for her infant
* Primary diagnosis in infant is unrelated to prematurity
* Infant not in legal and physical custody of the mother

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This is a study of first time biological mothers who, by definition, are female.
Enrollment: 208 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Maternal postpartum depression | The CESD-R will be administered at enrollment when the baby is approximately 2 days old
  Center for Epidemiological Studies Depression Scale-Revised (CESD-R). Scale is 0 - 36, where higher scores indicate higher levels of depressive symptoms.
Maternal postpartum depression | The CESD-R will be administered at 6 weeks
  Center for Epidemiological Studies Depression Scale-Revised (CESD-R). Scale is 0 - 36, where higher scores indicate higher levels of depressive symptoms.
Maternal postpartum depression | The CESD-R will be administered at 4 months
  Center for Epidemiological Studies Depression Scale-Revised (CESD-R). Scale is 0 - 36, where higher scores indicate higher levels of depressive symptoms.
Maternal parenting stress | The PSI-SF will be administered at enrollment when the baby is approximately 2 days old
  Parenting Stress Index-Short Form 4th Edition (PSI-SF). We will look at the Parental Distress subscale, which is interpreted based on percentile scores. Higher percentile scores indicate higher parental distress.
Maternal parenting stress | The PSI-SF will be administered at 6 weeks
  Parenting Stress Index-Short Form 4th Edition (PSI-SF). We will look at the Parental Distress subscale, which is interpreted based on percentile scores. Higher percentile scores indicate higher parental distress.
Maternal parenting stress | The PSI-SF will be administered at 4 months
  Parenting Stress Index-Short Form 4th Edition (PSI-SF)
Parenting confidence | The KPCS will be administered at 6 weeks
  The Karitane Parenting Confidence Scale (KPCS). The scale ranges from 0-45, with higher scores indicating higher confidence in parenting skills and abilities.
Parenting confidence | The KPCS will be administered at 4 months
  The Karitane Parenting Confidence Scale (KPCS). The scale ranges from 0-45, with higher scores indicating higher confidence in parenting skills and abilities.
Positive Parenting Quality | The WECS will be administered at 4 months
  Welch Emotional Connection Screen (WECS)

SECONDARY OUTCOMES:
Safe sleep practices | Infant care practices will be assessed at 6 weeks.
  Maternal report on questionnaire that child is put to sleep on their back, with no blankets, pillows, or other obstructions in the sleeping area.
Safe sleep practices | Infant care practices will be assessed at 4 months
  Maternal report on questionnaire that child is put to sleep on their back, with no blankets, pillows, or other obstructions in the sleeping area.
Breastfeeding | Infant care practices will be assessed at 6 weeks.
  Maternal report on questionnaire of feeding methods, including exclusive breastfeeding, formula supplement and short-term breastfeeding.
Breastfeeding | Infant care practices will be assessed at 4 months.
  Maternal report on questionnaire of feeding methods, including exclusive breastfeeding, formula supplement and any changes to feeding practices across first six weeks.
Participation in well child visits | Attendance at well child visits will be assessed at 4 months
  Maternal report on questionnaire of feeding methods, including exclusive breastfeeding, formula supplement and any changes to feeding practices across first 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Lise C Johnson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No